CLINICAL TRIAL: NCT04953637
Title: Combined Physiotherapy and Deep Brain Stimulation to Improve Independent Community Mobility in Parkinson's Disease
Brief Title: Physiotherapy and Deep Brain Stimulation in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor of Neurology, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-6338
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; deep brain stimulation; physiotherapy
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy group (Experimental): Participants assigned to the physiotherapy group will receive physiotherapy treatment at One Step Ahead Mobility physiotherapy clinic for 1-hour per day, 3 times/week for 8 weeks. They will begin to receive the physiotherapy treatment at 4 months following their surgery and once their DBS settings are optimized.
  Interventions: Other: Physiotherapy
- Control group (No Intervention): Participants assigned to the control group will not receive any additional intervention and will be precluded from starting formal physiotherapy for the duration of the study. However, they will be encouraged to keep an active lifestyle. In order to stay active, they will be recommended to do simple home exercises following a home exercise video that will be presented to them. They will be asked to do it 3 times/week for 8 weeks and keep an exercise log to help them stay on track.

INTERVENTIONS:
Other: Physiotherapy — Participants in the physiotherapy group will receive gait and balance focused physiotherapy at One Step Ahead Mobility physiotherapy clinic for 1-hour per day, 3 times/week for 8 weeks.
  Arms: Physiotherapy group

SUMMARY:
Deep brain stimulation (DBS) is the most commonly performed surgical treatment for individuals with Parkinson's disease (PD). DBS typically works best to lessen motor symptoms such as stiffness, slowness, and tremor. Despite an overall improvement of these motor symptoms with DBS, past research failed to show an increase in community mobility and have often reported an increase in falling after surgery. The ability to move around on one's own is important for functional independence and improved quality of life. There is growing evidence supporting the positive effects of physiotherapy on individuals with PD. Gait and balance training, in particular, can improve mobility and also prevent falls. So far, no study has shown the effectiveness of rehabilitation in patients receiving DBS.

The purpose of this study is to determine if DBS combined with physiotherapy is effective for improving safe independent mobility in individuals with PD, more so than with patients receiving DBS alone.

DETAILED DESCRIPTION:
This is a single-center, single-blind non-randomized controlled study, whereby individuals receiving DBS will be allocated to receive either physiotherapy or no intervention in keeping with current practice (control group).

Patients will be recruited from a pool of PD patients who have been identified as candidates for DBS in the Movement Disorders Clinics at the Toronto Western Hospital. Approximately 60 individuals will be recruited for the study. Study participation will span 8 months from the time of enrolment to the end of the study assessment.

Participants will be allocated to one of two groups: 1) physiotherapy, or 2) control. Participants living within 50 km of the physiotherapy clinic will be allocated to the physiotherapy group and those living beyond 50 km will be allocated to the control group. Participants assigned to the physiotherapy group will receive physiotherapy treatment at the One Step Ahead Mobility physiotherapy clinic for 1 hour per day, 3 times/week for 8 weeks. Participants assigned to the control group will not receive any additional intervention and will be precluded from starting formal physiotherapy for the duration of the study. However, they will be encouraged to keep an active lifestyle. In order to stay active, they will be recommended to do simple home exercises following a home exercise video that will be presented to them. Participants assigned to the control group will be assessed at the same points in time as participants in the physiotherapy group

All participants enrolled will undergo a similar timetable with assessments completed at five points throughout the study period. At month 0, participants are enrolled in the study, have their baseline assessment completed, and receive DBS surgery. At month 1, participants are started on optimization of DBS settings. At month 3, DBS settings are optimized and participants will have completed 7 days of activity monitoring using a wearable before the pre-intervention assessment. All participants are assessed before the physiotherapy group begins to receive gait and balance focused physiotherapy for 2 months (8 weeks) and the control group receives no intervention for 2 months. At month 5, physiotherapy is completed, and all participants undergo a third assessment immediately after the intervention period. At month 6, all participants are assessed with a Life Space Assessment questionnaire post-intervention and will have completed 7 days of activity monitoring using a wearable before the visit. At month 8, all participants undergo end of study assessment 3 months after completing physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* PD patients who have been identified as candidates for DBS.
* Ability to give informed consent.
* Patients ages 18 years and older.

Exclusion Criteria:

* Participants will be excluded if they have ongoing orthopaedic conditions potentially impacting on global mobility.
* Participants with severe cognitive deficits ((Montreal Cognitive Assessment (MoCA) score <17).
* Participants who are already receiving physiotherapy treatment (or that has been receiving it during the three months prior to enrollment) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mobility measures | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 4: Post-intervention assessment at month 6, and Visit 5: End of study assessment at month 8
  The primary outcome is the overall amount of independent mobility in the community. This will be measured with the Life Space Assessment (LSA) questionnaire. The LSA is a five-item questionnaire where participants are asked to indicate how often within the previous four weeks they moved within their homes, outside their homes but within their property, within their neighborhoods, within their towns, and outside their towns. LSA is a cross-sectional scale that quantifies the size of one's life space in the past 4 weeks as a score of 0-120 (0 = confined to the bedroom, 120 = daily travel to places outside of one's city/town).

SECONDARY OUTCOMES:
Balance | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  The Mini Balance Evaluation Systems Test (Mini-BESTest) will be used to measure dynamic balance. The Mini-BESTest is a 14-item test that includes four sections: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each item is scored from 0-2 (0 indicates that a person is unable to perform the task while a score of 2 is normal).
Gait | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Dynamic stability during walking, spatio-temporal gait variability and walking speed will be evaluated using the gait mat Zeno Walkway (ProtoKinetics, Havertown, PA, USA).
Balance confidence | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Balance confidence will be assessed using the Activity-specific Balance Confidence (ABC) scale. The ABC asks participants to rate, on a scale from 0-100%, how confident they would be performing 16 everyday tasks.
Number of falls and near falls | Collected over the 8 months' duration of the study and the diary will be reviewed at visits 2,3,4 and 5.
  Participants will be provided with a diary on enrolment into the study and will be asked to record any falls and near falls that they experience over the 8 months' duration of the study. A fall is defined as an event that result in a person coming to rest inadvertently on the ground or other lower level not due to a major intrinsic or extrinsic event. If a participant sustains a fall, they will be asked to record the details about the circumstances surrounding the fall with an open-ended questionnaire (setting, activity at the time of fall, physical injury, emergency department visit, hospitalization) in the falls diary. A near fall is defined as stumbling or loss of balance that would result in falling if sufficient recovery mechanisms were not activated. If the participant had a near fall, they will be asked to record the details about the event using the same open-ended questionnaire (setting, activity at the time of near fall, how the fall was avoided) in the diary.
Falls risk and functional mobility | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  The Timed Up and Go test (TUG) will be used to assess the falls risk and functional mobility. The TUG test is a physical performance measure in which the ability to rise up from a seated chair position, walk 3m, turn, walk back, and sit down is timed. The TUG test is highly correlated with functional mobility, gait speed, and falls in older adults.
Mood | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Mood will be assessed using the Beck Depression Inventory (BDI-I).The BDI-I is a 21-item questionnaire to assess depressive symptoms with a score of 0-3 for each item.
Anxiety | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  The Hamilton Anxiety Rate Scale (HAM-A) will be used to measure the anxiety symptoms. The scale consists of 14 items with a score of 0-4 for each item.
Exercise and activity levels | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Exercise and activity levels will be monitored through a set of questions about how much exercise or physical activity they do on a regularly. For the intensity of the activity, they will be asked to separate how much time they spend doing vigorous, moderate, and light activity.
Health-related quality of life | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Health-related quality of life will be assessed using the 39-item Parkinson's Disease Questionnaire (PDQ-39). The PDQ-39 asks participants to rate how often they encounter difficulty on items within eight subscales: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.
Parkinson's disease symptoms | Visit 1: Baseline assessment at month 0, Visit 2: Pre-intervention assessment at month 3, Visit 3: Post-intervention assessment at month 5, and Visit 5: End of study assessment at month 8
  Parkinson's disease symptoms will be evaluated with the Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) part 3 scores. The maximum total MDS-UPDRS score for part 3 ranges from 0 to 132. Higher scores indicate a worse outcome of Parkinson's disease.

OTHER OUTCOMES:
Exploratory outcome - average number of steps | 7 days of activity monitoring before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months
  A wearable activity monitor Fitbit Inspire 2 (Fitbit Inc., San Francisco, CA, USA) will be used to measure the average number of steps (the total number of steps per day averaged over the number of days worn). The participants will be provided with a Fitbit Inspire 2 activity monitor before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months. They will be instructed to wear the activity monitor on their wrist for 7 days including during sleep before the assessment visits.
Exploratory outcome - distance | 7 days of activity monitoring before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months
  A wearable activity monitor Fitbit Inspire 2 (Fitbit Inc., San Francisco, CA, USA) will be used to measure the distance (kilometers). The participants will be provided with a Fitbit Inspire 2 activity monitor before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months. They will be instructed to wear the activity monitor on their wrist for 7 days including during sleep before the assessment visits.
Exploratory outcome - physically active time | 7 days of activity monitoring before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months
  A wearable activity monitor Fitbit Inspire 2 (Fitbit Inc., San Francisco, CA, USA) will be used to measure the time being physically active. The participants will be provided with a Fitbit Inspire 2 activity monitor before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months. They will be instructed to wear the activity monitor on their wrist for 7 days including during sleep before the assessment visits.
Exploratory outcome - heart rate | 7 days of activity monitoring before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months
  A wearable activity monitor Fitbit Inspire 2 (Fitbit Inc., San Francisco, CA, USA) will be used to measure the heart rate (rates per minute). The participants will be provided with a Fitbit Inspire 2 activity monitor before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months. They will be instructed to wear the activity monitor on their wrist for 7 days including during sleep before the assessment visits.
Exploratory outcome - sleep quality | 7 days of activity monitoring before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months
  A wearable activity monitor Fitbit Inspire 2 (Fitbit Inc., San Francisco, CA, USA) will be used to measure sleep quality (minutes). The participants will be provided with a Fitbit Inspire 2 activity monitor before the pre-intervention assessment at 3 months and the post-intervention assessment at 6 months. They will be instructed to wear the activity monitor on their wrist for 7 days including during sleep before the assessment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fasano, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozano AM, Dostrovsky J, Chen R, Ashby P. Deep brain stimulation for Parkinson's disease: disrupting the disruption. Lancet Neurol. 2002 Aug;1(4):225-31. doi: 10.1016/s1474-4422(02)00101-1. PMID 12849455
- [Background] Kelly VE, Israel SM, Samii A, Slimp JC, Goodkin R, Shumway-Cook A. Assessing the effects of subthalamic nucleus stimulation on gait and mobility in people with Parkinson disease. Disabil Rehabil. 2010;32(11):929-36. doi: 10.3109/09638280903374139. PMID 19874214
- [Background] Yamada K, Goto S, Hamasaki T, Kuratsu JI. Effect of bilateral subthalamic nucleus stimulation on levodopa-unresponsive axial symptoms in Parkinson's disease. Acta Neurochir (Wien). 2008 Jan;150(1):15-22; discussion 22. doi: 10.1007/s00701-007-1451-3. Epub 2008 Jan 10. PMID 18180867
- [Background] Fasano A, Aquino CC, Krauss JK, Honey CR, Bloem BR. Axial disability and deep brain stimulation in patients with Parkinson disease. Nat Rev Neurol. 2015 Feb;11(2):98-110. doi: 10.1038/nrneurol.2014.252. Epub 2015 Jan 13. PMID 25582445
- [Background] Rochester L, Chastin SF, Lord S, Baker K, Burn DJ. Understanding the impact of deep brain stimulation on ambulatory activity in advanced Parkinson's disease. J Neurol. 2012 Jun;259(6):1081-6. doi: 10.1007/s00415-011-6301-9. Epub 2011 Nov 16. PMID 22086738
- [Background] Daneault JF, Duval C, Barbat-Artigas S, Aubertin-Leheudre M, Jodoin N, Panisset M, Sadikot AF. Subthalamic stimulation improves motor function but not home and neighborhood mobility. Mov Disord. 2014 Dec;29(14):1816-9. doi: 10.1002/mds.25911. Epub 2014 May 22. PMID 24849309
- [Background] Tudor-Locke C, Craig CL, Aoyagi Y, Bell RC, Croteau KA, De Bourdeaudhuij I, Ewald B, Gardner AW, Hatano Y, Lutes LD, Matsudo SM, Ramirez-Marrero FA, Rogers LQ, Rowe DA, Schmidt MD, Tully MA, Blair SN. How many steps/day are enough? For older adults and special populations. Int J Behav Nutr Phys Act. 2011 Jul 28;8:80. doi: 10.1186/1479-5868-8-80. PMID 21798044
- [Background] Allert N, Cheeran B, Deuschl G, Barbe MT, Csoti I, Ebke M, Glaser M, Kang JS, Kelm S, Krack P, Kroth J, Jobst U, Leisse M, Oliviero A, Nolte PN, Quick-Weller J, Strothjohann M, Tamas G, Werner M, Muthuraman M, Volkmann J, Fasano A, Groppa S. Postoperative rehabilitation after deep brain stimulation surgery for movement disorders. Clin Neurophysiol. 2018 Mar;129(3):592-601. doi: 10.1016/j.clinph.2017.12.035. Epub 2018 Jan 10. PMID 29414403
- [Background] Tomlinson CL, Patel S, Meek C, Herd CP, Clarke CE, Stowe R, Shah L, Sackley C, Deane KH, Wheatley K, Ives N. Physiotherapy intervention in Parkinson's disease: systematic review and meta-analysis. BMJ. 2012 Aug 6;345:e5004. doi: 10.1136/bmj.e5004. PMID 22867913
- [Background] Tomlinson CL, Patel S, Meek C, Herd CP, Clarke CE, Stowe R, Shah L, Sackley CM, Deane KH, Wheatley K, Ives N. Physiotherapy versus placebo or no intervention in Parkinson's disease. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD002817. doi: 10.1002/14651858.CD002817.pub4. PMID 24018704
- [Background] Smania N, Corato E, Tinazzi M, Stanzani C, Fiaschi A, Girardi P, Gandolfi M. Effect of balance training on postural instability in patients with idiopathic Parkinson's disease. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):826-34. doi: 10.1177/1545968310376057. PMID 21045119
- [Background] Shen X, Mak MK. Repetitive step training with preparatory signals improves stability limits in patients with Parkinson's disease. J Rehabil Med. 2012 Nov;44(11):944-9. doi: 10.2340/16501977-1056. PMID 23027184
- [Background] Shen X, Mak MK. Technology-assisted balance and gait training reduces falls in patients with Parkinson's disease: a randomized controlled trial with 12-month follow-up. Neurorehabil Neural Repair. 2015 Feb;29(2):103-11. doi: 10.1177/1545968314537559. Epub 2014 Jun 24. PMID 24961993
- [Background] Ferrazzoli D, Ortelli P, Madeo G, Giladi N, Petzinger GM, Frazzitta G. Basal ganglia and beyond: The interplay between motor and cognitive aspects in Parkinson's disease rehabilitation. Neurosci Biobehav Rev. 2018 Jul;90:294-308. doi: 10.1016/j.neubiorev.2018.05.007. Epub 2018 May 4. PMID 29733882
- [Background] Grobbelaar R, Venter R, Welman KE. Backward compared to forward over ground gait retraining have additional benefits for gait in individuals with mild to moderate Parkinson's disease: A randomized controlled trial. Gait Posture. 2017 Oct;58:294-299. doi: 10.1016/j.gaitpost.2017.08.019. Epub 2017 Aug 18. PMID 28843186
- [Background] Baker PS, Bodner EV, Allman RM. Measuring life-space mobility in community-dwelling older adults. J Am Geriatr Soc. 2003 Nov;51(11):1610-4. doi: 10.1046/j.1532-5415.2003.51512.x. PMID 14687391
- [Background] Zhu L, Duval C, Boissy P, Montero-Odasso M, Zou G, Jog M, Speechley M. Comparing GPS-Based Community Mobility Measures with Self-report Assessments in Older Adults with Parkinson's Disease. J Gerontol A Biol Sci Med Sci. 2020 Nov 13;75(12):2361-2370. doi: 10.1093/gerona/glaa012. PMID 31957792
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Leddy AL, Crowner BE, Earhart GM. Utility of the Mini-BESTest, BESTest, and BESTest sections for balance assessments in individuals with Parkinson disease. J Neurol Phys Ther. 2011 Jun;35(2):90-7. doi: 10.1097/NPT.0b013e31821a620c. PMID 21934364
- [Background] Steffen T, Seney M. Test-retest reliability and minimal detectable change on balance and ambulation tests, the 36-item short-form health survey, and the unified Parkinson disease rating scale in people with parkinsonism. Phys Ther. 2008 Jun;88(6):733-46. doi: 10.2522/ptj.20070214. Epub 2008 Mar 20. Erratum In: Phys Ther. 2010 Mar;90(3):462. PMID 18356292
- [Background] The prevention of falls in later life. A report of the Kellogg International Work Group on the Prevention of Falls by the Elderly. Dan Med Bull. 1987 Apr;34 Suppl 4:1-24. PMID 3595217
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Pohl P, Nordin E, Lundquist A, Bergstrom U, Lundin-Olsson L. Community-dwelling older people with an injurious fall are likely to sustain new injurious falls within 5 years--a prospective long-term follow-up study. BMC Geriatr. 2014 Nov 18;14:120. doi: 10.1186/1471-2318-14-120. PMID 25407714
- [Background] Stack E, Ashburn A. Fall events described by people with Parkinson's disease: implications for clinical interviewing and the research agenda. Physiother Res Int. 1999;4(3):190-200. doi: 10.1002/pri.165. PMID 10581625
- [Background] Gazibara T, Kisic Tepavcevic D, Svetel M, Tomic A, Stankovic I, Kostic VS, Pekmezovic T. Near-falls in people with Parkinson's disease: Circumstances, contributing factors and association with falling. Clin Neurol Neurosurg. 2017 Oct;161:51-55. doi: 10.1016/j.clineuro.2017.08.008. Epub 2017 Aug 24. PMID 28858631
- [Background] Lindholm B, Hagell P, Hansson O, Nilsson MH. Prediction of falls and/or near falls in people with mild Parkinson's disease. PLoS One. 2015 Jan 30;10(1):e0117018. doi: 10.1371/journal.pone.0117018. eCollection 2015. PMID 25635687
- [Background] Nocera JR, Stegemoller EL, Malaty IA, Okun MS, Marsiske M, Hass CJ; National Parkinson Foundation Quality Improvement Initiative Investigators. Using the Timed Up & Go test in a clinical setting to predict falling in Parkinson's disease. Arch Phys Med Rehabil. 2013 Jul;94(7):1300-5. doi: 10.1016/j.apmr.2013.02.020. Epub 2013 Mar 6. PMID 23473700
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Pradhan S, Kelly VE. Quantifying physical activity in early Parkinson disease using a commercial activity monitor. Parkinsonism Relat Disord. 2019 Sep;66:171-175. doi: 10.1016/j.parkreldis.2019.08.001. Epub 2019 Aug 3. PMID 31420310
- [Background] Lamont RM, Daniel HL, Payne CL, Brauer SG. Accuracy of wearable physical activity trackers in people with Parkinson's disease. Gait Posture. 2018 Jun;63:104-108. doi: 10.1016/j.gaitpost.2018.04.034. Epub 2018 Apr 24. PMID 29729611